CLINICAL TRIAL: NCT00252343
Title: An Eight-Week, Double-Blind, Placebo-Controlled, Multicenter Study With Escitalopram (10mg qd) as Positive Control, Evaluating the Efficacy, Safety, Tolerability of a Fixed Dose of SR58611A (350 mg q12) in Outpatients With Generalized Anxiety Disorder
Brief Title: Efficacy and Safety of SR58611A in Patients With a Generalized Anxiety Disorder
Acronym: LIBRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5892
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Anxiety Disorder
Keywords: anxiety disorder
MeSH Terms: conditions — Anxiety Disorders | interventions — Amibegron hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SR58611A

SUMMARY:
To evaluate the efficacy of a fixed dose of SR58611A (350mg q12) compared to placebo in patients with GeneralizedAnxiety Disorder (GAD) using escitalopram (10 mg qd) as positive control. To evaluate the tolerability and safety of SR58611A in patients with GAD.

DETAILED DESCRIPTION:
The current study will be conducted to evaluate the efficacy, safety, and tolerability of SR58611A (350 mg q12) compared to placebo in patients with generalized anxiety disorder (GAD), using escitalopram (10 mg qd) as a positive control. This is an 8-week, double-blind, randomized, 3-parallel-group, placebo- and escitalopram-controlled, study.A 1-week, placebo, single-blind period precedes the 8-week randomized treatment period. A Safety Follow up Visit (Segment C) is scheduled 1 week after the acute treatmentperiod (Segment B) or early termination. This trial is designed to compare the efficacy, safety, and tolerability of SR58611A to placebo. In this study, escitalopram, a selective serotonin reuptake inhibitor (SSRI) antidepressant, is used as a positive control and has been chosen as the comparator agentas it is approved for treatment of GAD at a dose of 10 mg once daily.

ELIGIBILITY:
Inclusion Criteria:

Main inclusion criteria:

1. Out-patients, 18 year and older.
2. Generalized Anxiety Disorder (GAD) according toDSM-IV-TR criteria / MINI.
3. Minimum total score of 20 on the 14-item HamiltonAnxiety Rating Scale (HAM-A)

Exclusion Criteria:

Main exclusion criteria:

1. Patients with a diagnosis of Major Depressive Disorder within 6 months of study entry.
2. Patients with a Montgomery-Asberg Depression Rating Scale (MADRS) total score of 18 or higher
3. Patients who are assessed to have a moderate to high current risk for suicide according to the MINI, or at imminent risk for a suicide attempt
4. Patients with other current anxiety disorder (within 6 months) assessed with the MINI:- Agoraphobia, social phobia,- Panic disorder,- Obsessive compulsive disorder,- Post-traumatic stress disorder, acute stress disorder.
5. Patients with a lifetime history according to the MINI of:- Bipolar disorders,- Psychotic disorders,- Antisocial Personality Disorder.
6. Patients with a current history according to the MINI of:- Anorexia nervosa or bulimia nervosa in the past 6 months,- Alcohol dependence or abuse or substance dependence or abuse in the past 12 months except nicotine or caffeine dependence.
7. Patients who have received non-pharmacologic, somatic treatments for psychiatric disease
8. Patients who have initiated, stopped, or changed the frequency or nature of psychotherapy within 3 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2005-09; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
14-item Hamilton Anxiety Rating Scale (HAM-A) total score

SECONDARY OUTCOMES:
Change from baseline in Clinical Global Impression (CGI)
Severity of Illness score
Safety assessments

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com